CLINICAL TRIAL: NCT07360925
Title: Direct Measurement of Pericoronary Adipocyte Size Gradient as a Parameter of Immunometabolic Changes of Perivascular Adipose Tissue
Brief Title: Pericoronary Adipocyte Size Gradient
Acronym: AdipoCor
Status: Recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Ivana Kralova Lesna, Ivana Kralova Lesna, M.D., PhD., assoc. prof., Institute for Clinical and Experimental Medicine
Other Study IDs: AdipoCor2023
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Heart Transplantation
Keywords: Pericoronary adipose tissue; adipocyte size; inflammatory changes; macrophages
MeSH Terms: conditions — Heart Failure | interventions — Heart Transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Coronary artery segment with adjacent tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- patients with advanced heart failure: A group of patients with advanced heart failure were indicated for heart transplanta-tion for either ischemic or dilatational cardiomyopathy. The study group will also in-clude subjects with previously implanted LVAD as a bridge-to-transplant approach. Predictory-related subgroups will be evaluated separately.
  Interventions: Procedure: Heart transplantation for the final stage of heart failure

INTERVENTIONS:
Procedure: Heart transplantation for the final stage of heart failure — The study population comprises patients who underwent heart transplantation for heart failure at the Institute for Clinical and Experimental Medicine, Cardiovascular Surgery Department, between June 2023 and December 2028. Only the subjects' retrospective clinical data and matching heart samples will be analyzed.

SUMMARY:
Evaluation of pericoronary adipocyte gradient (PCAT) in relationship with local atherosclerotic changes in a patient undergoing heart transplantation.

DETAILED DESCRIPTION:
The project is designed to analyze the impact of inflammation spreading from pericoro-nary adipose tissue to the arterial wall or vice versa. Adipocyte size and immunometabolic parameters gradients established from independent analysis of samples closely adjacent to the coronary artery and those more distant from the arterial lumen will be used to establish the direction of inflammation propagation. The coronary arteries, along with adjacent pericoronary adipose tissue, from explanted hearts will be obtained during heart transplantation of patients with advanced atherosclerosis (ischemic heart disease) and with less advanced atherosclerotic disease (dilated cardiomyopathy).

Clinical data (including age, BMI, comorbidities, and concomitant medications) will be recorded. Specifically, previous left ventricular assist device (LVAD) implantation, used as a bridge-to-transplant approach, will be followed to establish the effect of artificial hemodynamic disturbance on coronary artery blood flow on study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-90 years
* Diagnosis of dilatational or ischemic cardiomyopathy
* Patients undergoing heart transplantation in IKEM

Exclusion Criteria:

* Known combined diagnosis of dilatational and ischemic cardiomyopathy
* Arrhythmogenic cardiomyopathy
* Congenital heart defects
* Non-eligibility due to the absence of informed consent

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients who underwent heart transplantation for heart failure at the Institute for Clinical and Experimental Medicine, Cardiovascular Surgery Department, between June 2023 and December 2028. Only the subjects' ret-rospective clinical data and matching heart samples will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Adipocyte size | Perioperative/Periprocedural
  Assessment of the difference (in square micrometer) between adipocyte size closely adjacent to the coronary artery and those more distant from the arterial lumen in relation to atherosclerotic pathologies in situ

SECONDARY OUTCOMES:
Immunological parameters | Perioperative/Periprocedural
  The immunological characteristics-T cells (counts and percentages), B cells (counts and percentages), macrophages and their subpopulations (counts and percentages)-and the immunohistochemical biomarkers sclerostin, TREM-2 (triggering receptor expressed on myeloid cells 2), and mimecan (score) in the arterial wall and pericoronary adipose tissue (PCAT) will be analyzed and compared.
Morphological parameters | Perioperative/Periprocedural
  The morphological characteristics-atherosclerotic plaque type (category) and calcification rate (percentage)-in the arterial wall and pericoronary adipose tissue (PCAT) will be analyzed and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Experimental Medicine, Institute for Clinical and Experimental Medicine,, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No